CLINICAL TRIAL: NCT03513913
Title: Comparison of the Effect of Conventional IVF and ICSI Fertilization Method on Human IVF Treatment Outcome
Brief Title: Comparison of IVF and ICSI in Human IVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Peter Fancsovits, Ph.D., Senior cilincal embryologyst, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SemmelweisU-003
Record Dates: First submitted 2018-03-26; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Infertility
Keywords: in vitro fertilization; intracytoplasmic sperm injection; fertilization; Assisted reproduction
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVF (Experimental): Oocytes fertilized by conventional in vitro fertilization (IVF) method
  Interventions: Procedure: ICSI
- ICSI (Experimental): Oocytes fertilized by intracytoplasmic sperm injection (ICSI) method
  Interventions: Procedure: ICSI

INTERVENTIONS:
Procedure: ICSI — Oocytes are fertilized by conventional in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI)

SUMMARY:
In this prospective randomized clinical trial we plan to compare two fertilization method which are widely used during in vitro fertilization (IVF) treatment. Outcome of conventional IVF and intracytoplasmic sperm injection (ICSI) treatment will be compared in this study.

ELIGIBILITY:
Inclusion Criteria:

Infertile patients entering in vitro fertilization treatment At least 1 oocytes collected Semen sample is suitable for IVF and ICSI fertilization as well Number of oocytes collected is lower than 5 AND/OR female age is equal or more than 40 years

Exclusion Criteria:

Samen sample is not suitable for conventional IVF fertilization Previous conventional IVF treatment resulted in <50% fertilization rate

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-04-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Fertilization rate | 18 hours after insemination
  Number of oocytes fertilized

SECONDARY OUTCOMES:
Embryo quality | 36 and 72 hours after fertilization
  Number and quality of blastomeres, amount of fragmentation, embryo grade
Implantation rate | 4 weeks after embryo transfer
  Number of embryos implanted (/number of embryos transferred)
Clinical pregnancy rate | 4 weeks after the embryo transfer
  Number of clinical pregnancies (/No. of embryo transfers)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fancsovits, PhD, Study Chair — Semmelweis University First Department of Obstetrics and Gynecology, Budapest, Hungary; Janos Urbancsek, DSc, Principal Investigator — Semmelweis University First Department of Obstetrics and Gynecology, Budapest, Hungary; Csaba Pribenszky, PhD, Principal Investigator — University of Veterinary Science, Budapest, Hungary; Adam Lehner, PhD, Principal Investigator — Semmelweis University First Department of Obstetrics and Gynecology, Budapest, Hungary; Zita Kaszás, BSc, Principal Investigator — Semmelweis University First Department of Obstetrics and Gynecology, Budapest, Hungary; Miklós I Ács, MD, Principal Investigator — Klinikum Kempten Oberallgäu, Kempten, Germany
Locations (1):
- Semmelweis University First Department of Obstetrics and Gynecology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No